CLINICAL TRIAL: NCT03932071
Title: The Efficacy of New Adjuvant Chemotherapy of Osteosarcoma Combined With Zoledronic Acid in Decrease the Lung Metastatic Rate of Osteosarcoma
Brief Title: Zoledronic Acid in Decrease the Lung Metastatic Rate of Osteosarcoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhaoming Ye, Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChiCTR-IPR-16008568
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Lung Metastases; Tumor Necrosis
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- experimental group (Experimental)
  Interventions: Drug: Zoledronic Acid
- control group (No Intervention)

INTERVENTIONS:
Drug: Zoledronic Acid
  Arms: experimental group

SUMMARY:
Zoledronic acid is an adjuvant treatment for primary osteosarcoma. Zoledronic acid has been widely used in the treatment of metastatic bone tumors. In addition to its inhibition of tumor osteoclasis, it also produces certain killing of tumor cells. effect. Foreign studies have shown that zoledronic acid also has a killing effect on osteosarcoma and has a certain inhibitory effect on distant metastasis. We hope that it can reduce tumor recurrence and lung metastasis through this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteosarcoma who were diagnosed with initial pathology and pathology were excluded from lung metastasis or other metastatic lesions by CT and total body emission-computed tomography, and patients with standard chemotherapy were evaluated.

Exclusion Criteria:

* Pulmonary metastasis, pregnancy or lactation, renal insufficiency (creatinine clearance <70 ml/min/1.73 m2), liver dysfunction, obvious oral disease, and unsuitable for bisphosphonate treatment after evaluation, have been found. With diseases that still require hormone therapy, abnormal blood system, heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
rate of lung metastasis | 3 year
  Discovery the rate of neonatal lung metastases by high-resolution chest CT
rate of tumor recurrence | 3 year
  Local recurrence rate of tumor or rate of distant metastasis

SECONDARY OUTCOMES:
rate of tumor necrosis less than 90% | 3 year
  the rate of patients that postoperative tumor necrosis rate was estimated to be lower than grade III（90%）

CONTACTS AND LOCATIONS:
Overall Officials: zhaoming Ye, Prof., Principal Investigator — 2nd Affiliated Hospital Of Zhejiang University
Locations (1):
- 2nd Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No